CLINICAL TRIAL: NCT07192003
Title: Comparison of the Immediate Effect of Flossband and Mobilization With Movement on Shoulder Mobility in Volleyball Athletes: A Randomized Clinical Trial
Brief Title: Immediate Effects of Flossband and Mobilization With Movement on Shoulder Mobility in Volleyball Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Valéria Mayaly Alves de Oliveira, Professor, Researcher, and Principal Investigator (PhD), Federal University of Paraíba, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 7812025
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy Athlete; Shoulder Mobility; Musculoskeletal Health
Keywords: Range of Motion; Shoulder; Sports; Physical Therapy Modalities; Mobilization with Movement; Volleyball
MeSH Terms: interventions — Movement; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with Movement (MWM) Group (Active Comparator): Participants in this arm will perform the standardized Mobilization with Movement (MWM) protocol. While seated in a chair with back support and hips, knees, and ankles at 90° flexion, the researcher will stabilize the scapula with one hand and apply a posterolateral glide to the anterior humeral head with the other hand during active shoulder elevation in the scapular plane. The intervention consists of 3 sets of 10 repetitions, with a 1-minute rest interval between sets. Assessments will be conducted at baseline and immediately post-intervention, including shoulder range of motion using a digital inclinometer, perception of movement fluency using a Visual Analogue Scale (VAS), and sport-specific performance tests (One-arm Seated Shot Put Test and Functional Throwing Performance Index).
  Interventions: Other: Mobilization with Movement (MWM) Group
- Floss Band Group (FBG) (Experimental): Participants in this arm will perform the standardized Floss Band (FBG) protocol. While seated with the shoulder at 90° abduction, the researcher will apply a compressive elastic band made of 100% polymer gel (T.P.E), measuring 210 cm in length, 5 cm in width, and 1.3 mm in thickness. The first anchor is placed two fingers medial to the acromion, and the band is wrapped around the shoulder until the second anchor at the end of the band is fixed. After the application, the participant will perform sport-specific movements (spike and serve) for 2 minutes. Following the completion of the compression period, the band will be removed. Assessments will be conducted at baseline and immediately post-intervention, including shoulder range of motion using a digital inclinometer, perception of movement fluency using a Visual Analogue Scale (VAS), and sport-specific performance tests (One-arm Seated Shot Put Test and Functional Throwing Performance Index).
  Interventions: Device: Floss Band Group (FBG)

INTERVENTIONS:
Device: Floss Band Group (FBG) — Participants in this arm will perform the standardized Floss Band (FBG) protocol. While seated with the shoulder at 90° abduction, the researcher will apply a compressive elastic band made of 100% polymer gel (T.P.E), measuring 210 cm in length, 5 cm in width, and 1.3 mm in thickness. The first anchor is placed two fingers medial to the acromion, and the band is wrapped around the shoulder until the second anchor at the end of the band is fixed. After the application, the participant will perform sport-specific movements (spike and serve) for 2 minutes. Following the completion of the compression period, the band will be removed. Assessments will be conducted at baseline and immediately post-intervention, including shoulder range of motion using a digital inclinometer, perception of movement fluency using a Visual Analogue Scale (VAS), and sport-specific performance tests (One-arm Seated Shot Put Test and Functional Throwing Performance Index).
  Arms: Floss Band Group (FBG)
Other: Mobilization with Movement (MWM) Group — Participants in this arm will perform the standardized Mobilization with Movement (MWM) protocol. While seated in a chair with back support and hips, knees, and ankles at 90° flexion, the researcher will stabilize the scapula with one hand and apply a posterolateral glide to the anterior humeral head with the other hand during active shoulder elevation in the scapular plane. The intervention consists of 3 sets of 10 repetitions, with a 1-minute rest interval between sets. Assessments will be conducted at baseline and immediately post-intervention, including shoulder range of motion using a digital inclinometer, perception of movement fluency using a Visual Analogue Scale (VAS), and sport-specific performance tests (One-arm Seated Shot Put Test and Functional Throwing Performance Index).
  Arms: Mobilization with Movement (MWM) Group

SUMMARY:
The goal of this clinical trial is to learn if Floss Band application works as effectively as mobilization with movement (MWM) to improve shoulder mobility in volleyball athletes. It will also explore whether these techniques affect athletes' perception of movement fluency and sport-specific performance.

The main questions it aims to answer are:

Does Floss Band application immediately improve shoulder range of motion in volleyball athletes? Does Floss Band application change the perception of movement fluency compared to MWM? Does Floss Band application impact sport-specific performance tests compared to MWM?

Participants will:

Be randomly assigned to receive either Floss Band or mobilization with movement Have their shoulder mobility, perception of movement, and sport performance tested before and immediately after the intervention

DETAILED DESCRIPTION:
Overhead sports such as volleyball demand repetitive, high-velocity arm movements that predispose athletes to musculoskeletal adaptations, especially in the glenohumeral joint. Among these, glenohumeral internal rotation deficit (GIRD) is a frequent finding, typically associated with posterior capsular tightness and muscular adaptations. This condition has been linked to decreased shoulder performance and a greater risk of overuse injuries.

Conservative approaches are essential for preserving mobility and reducing injury risk in overhead athletes. Mobilization with movement (MWM) is a well-established manual therapy intervention, combining therapist-applied accessory glenohumeral mobilization with the athlete's active shoulder motion. Evidence supports its capacity to produce immediate improvements in range of motion and sensorimotor control.

In contrast, the use of compressive elastic bands, or Floss Bands, represents a more recent strategy in rehabilitation. Proposed mechanisms include transient ischemia followed by reperfusion, improved soft tissue gliding, neuromuscular activation, and increased proprioceptive input. Although Floss Band applications have gained popularity, robust evidence on their effects in overhead athletes is still limited.

The current randomized, controlled, double-blind equivalence trial aims to compare the immediate effects of Floss Band application with MWM on shoulder mobility in volleyball athletes. The equivalence design was selected because both interventions are hypothesized to provide similar clinical benefits, and the study seeks to determine whether the novel approach (Floss Band) is not inferior to the well-established MWM.

Intervention Procedures Participants will undergo two assessments: baseline and immediately post-intervention. Interventions will be delivered by researchers trained and standardized in both techniques.

Floss Band Group (FBG): The participant will be seated with the shoulder positioned at 90° abduction. The researcher will apply a compressive elastic band (100% polymer gel, 210 cm circumference, 5 cm width, 1.3 mm thickness). The first anchor will be placed two finger-widths medial to the acromion, and the band will be wrapped circumferentially around the shoulder until the material length is exhausted, securing the final anchor. During the two-minute application, the participant will perform sport-specific movements (e.g., spike and serve gestures). After the time limit, the band will be removed.

Mobilization with Movement Group (MWM): The participant will remain seated with back support and hips, knees, and ankles flexed at 90°. The therapist will stabilize the scapula with one hand, while the other hand will apply a posterolateral glide to the humeral head during active arm elevation in the scapular plane. The protocol will consist of three sets of 10 repetitions, with one-minute rest intervals between sets.

Data Management and Quality Assurance All assessors will undergo standardized training to ensure consistency across evaluations. Prior to trial initiation, pilot testing of procedures will be conducted. Data will be collected using predefined case report forms and transferred into a secure electronic database.

Quality assurance measures will include:

Data validation: Automated checks for range, completeness, and logical consistency between variables.

Source data verification: Cross-checks of electronic entries with original case report forms by an independent monitor.

Auditing: Periodic audits conducted by external staff not involved in data collection or intervention delivery.

Standard Operating Procedures (SOPs): Detailed instructions for participant recruitment, intervention delivery, data entry, adverse event reporting, and change management.

Data dictionary: Comprehensive description of variables, coding schemes, and reference values to maintain consistency and transparency.

Sample Size and Statistical Plan The trial is powered to detect equivalence between interventions in the primary outcome (shoulder ROM). A total of 36 athletes will be randomized equally across groups, stratified by sex and age. Analyses will follow the intention-to-treat principle. Between-group differences will be adjusted for baseline values, and 95% confidence intervals will be calculated to test equivalence margins. Missing data will be addressed with multiple imputation methods.

Expected Contribution By comparing an innovative compressive technique with an established manual therapy, this study is designed to provide high-quality evidence on immediate intervention effects in volleyball athletes. The results are expected to inform clinicians, coaches, and sports medicine professionals on effective strategies for optimizing shoulder function and preventing injury in overhead sports.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Male or female volleyball athletes (indoor or beach), at amateur or professional level.
* Regular training routine of at least two sessions per week.
* No shoulder pain at the time of testing or during the previous three months.

Exclusion Criteria:

* History of shoulder surgery, structural shoulder injuries (e.g., fractures, labrum tear), or recurrent glenohumeral dislocation.
* Skin disorders contraindicating the intervention, including active dermatitis, inflammatory-phase psoriasis, cutaneous infections (e.g., folliculitis), open wounds, burns, eczema, or hypersensitivity in the shoulder region.
* Vascular disorders contraindicating the intervention, including history or diagnosis of deep vein thrombosis, symptomatic varicose veins, peripheral arterial disease, lymphedema, or advanced chronic venous insufficiency.
* Other conditions contraindicating intervention: peripheral neuropathies with significant sensory loss, presence of a pacemaker in the region of band application, known allergy to elastic band material, or pain during shoulder movement at assessment.
* Development of shoulder or elbow injuries during the study, especially requiring surgical intervention.
* Participants who voluntarily withdraw from the study at any time.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Motion - External Rotation | Baseline (prior to intervention, Day 1) and post-intervention (Day 1)
  Glenohumeral external rotation (dominant shoulder) will be measured using the Baseline® Digital Inclinometer. The participant will lie in the supine position with the shoulder abducted to 90°, elbow flexed to 90°, and forearm in neutral. The inclinometer will be placed on the anterior mid-forearm, and the participant will perform active external rotation. Three measurements will be taken, and the mean value will be calculated for analysis.
Shoulder Range of Motion - Internal Rotation, Flexion, Abduction, Horizontal Abduction | Baseline (prior to intervention, Day 1) and post-intervention (Day 1)
  Internal rotation: same supine position, inclinometer on posterior mid-forearm.
  Flexion and abduction: seated with hips, knees, and ankles at 90° flexion; inclinometer on anterior humerus for flexion, lateral mid-humerus for abduction.
  Horizontal abduction: supine, shoulder 90° abduction, 90° external rotation, elbow 90° flexion; inclinometer on anterior mid-humerus.
  Three measurements per movement will be recorded and averaged.

SECONDARY OUTCOMES:
Functional Performance - One-arm Seated Single Arm Shot Put Test (OSP) | Baseline (prior to intervention, Day 1) and post-intervention (Day 1)
  Participants will be seated with back against a wall, knees flexed, feet on the floor. The non-tested arm will be positioned on the chest or alongside the body. Participants will throw a 3kg medicine ball overhead, simulating a spike/serve, over a 10 m marked distance. Two submaximal familiarization trials will be performed, followed by three attempts with 1-minute rest intervals. The mean distance of the three attempts will be calculated.
Functional Throwing Performance Index (FTPI) | Baseline (prior to intervention, Day 1) and post-intervention (Day 1)
  Participants will stand 4.6 meters from a 30.5 × 30.5 cm target on a wall at 1.22 m height. Using a rubber ball (~50.8 cm circumference), participants will throw toward the target, catch the rebound, and repeat for three 30-second trials. Eight warm-up throws will be performed prior. FTPI = number of successful hits ÷ total throws.
Perceived Movement Fluency (VAS) | Immediately post-intervention (Day 1)
  Participants will rate their subjective perception of shoulder movement fluency during spike/serve on a 10 cm visual analogue scale (0 = "stiff/irregular movement," 10 = "completely fluid/smooth"). The distance from the left end of the line to the participant's mark will be recorded as the final score.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba, Igarapé-Açu, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected in this study, including de-identified measurements of shoulder range of motion, functional performance tests, and perceived movement fluency, will be made available to other researchers. Data dictionaries describing each variable, coding, and units will also be provided. Sharing will occur in accordance with participant consent, ethical approvals, and data privacy regulations, after the publication of the main study results.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be made available starting 6 months after publication of the main study results and will remain accessible for 5 years.
Access Criteria: Data will be shared with qualified researchers upon request. Researchers must submit a data access request and sign a data use agreement outlining the intended analyses and ensuring confidentiality. Requests will be reviewed by the principal investigator to ensure that proposed use aligns with the study objectives and ethical standards.

REFERENCES:
- [Background] Young WK, Briner W, Dines DM. Epidemiology of Common Injuries in the Volleyball Athlete. Curr Rev Musculoskelet Med. 2023 Jun;16(6):229-234. doi: 10.1007/s12178-023-09826-2. Epub 2023 Apr 4. PMID 37014607
- [Background] Wassinger CA, Myers JB, Gatti JM, Conley KM, Lephart SM. Proprioception and throwing accuracy in the dominant shoulder after cryotherapy. J Athl Train. 2007 Jan-Mar;42(1):84-9. PMID 17597948
- [Background] Wang S, Zeng J, Mani R, Chapple CM, Ribeiro DC. The immediate effects of mobilization with movement on shoulder range of motion and pain in patients with rotator cuff-related shoulder pain: A randomized controlled trial (Evolution Trial). Braz J Phys Ther. 2024 Nov-Dec;28(6):101145. doi: 10.1016/j.bjpt.2024.101145. Epub 2024 Nov 20. PMID 39571379
- [Background] Tozzo MC, Ansanello W, Martins J, Zatiti SCA, de Oliveira AS. Inclinometer Reliability for Shoulder Ranges of Motion in Individuals With Subacromial Impingement Syndrome. J Manipulative Physiol Ther. 2021 Mar;44(3):236-243. doi: 10.1016/j.jmpt.2020.12.001. Epub 2021 Apr 27. PMID 33926742
- [Background] Tooth C, Gofflot A, Schwartz C, Croisier JL, Beaudart C, Bruyere O, Forthomme B. Risk Factors of Overuse Shoulder Injuries in Overhead Athletes: A Systematic Review. Sports Health. 2020 Sep/Oct;12(5):478-487. doi: 10.1177/1941738120931764. Epub 2020 Aug 6. PMID 32758080
- [Background] Tagliarini GO, Junior JRS, Barbosa GMP, Secchi LLB. Performance, Test-retest Reliability, and Measurement Error of the Upper Limb Seated Shot Put Test According to Different Positions of Execution. Int J Sports Phys Ther. 2023 Jun 1;V18(3):698-706. doi: 10.26603/001c.75227. eCollection 2023. PMID 37425121
- [Background] Schwank A, Blazey P, Asker M, Moller M, Hagglund M, Gard S, Skazalski C, Haugsbo Andersson S, Horsley I, Whiteley R, Cools AM, Bizzini M, Ardern CL. 2022 Bern Consensus Statement on Shoulder Injury Prevention, Rehabilitation, and Return to Sport for Athletes at All Participation Levels. J Orthop Sports Phys Ther. 2022 Jan;52(1):11-28. doi: 10.2519/jospt.2022.10952. PMID 34972489
- [Background] Satpute K, Reid S, Mitchell T, Mackay G, Hall T. Efficacy of mobilization with movement (MWM) for shoulder conditions: a systematic review and meta-analysis. J Man Manip Ther. 2022 Feb;30(1):13-32. doi: 10.1080/10669817.2021.1955181. Epub 2021 Aug 1. PMID 34334099
- [Background] Rose MB, Noonan T. Glenohumeral internal rotation deficit in throwing athletes: current perspectives. Open Access J Sports Med. 2018 Mar 19;9:69-78. doi: 10.2147/OAJSM.S138975. eCollection 2018. PMID 29593438
- [Background] Pascoal AG, Ribeiro A, Infante J. Scapular Resting Posture and Scapulohumeral Rhythm Adaptations in Volleyball Players: Implications for Clinical Shoulder Assessment in Athletes. Sports (Basel). 2023 Jun 8;11(6):114. doi: 10.3390/sports11060114. PMID 37368564
- [Background] Myers JB, Oyama S, Goerger BM, Rucinski TJ, Blackburn JT, Creighton RA. Influence of humeral torsion on interpretation of posterior shoulder tightness measures in overhead athletes. Clin J Sport Med. 2009 Sep;19(5):366-71. doi: 10.1097/JSM.0b013e3181b544f6. PMID 19741307
- [Background] Mine K, Nakayama T, Milanese S, Grimmer K. Effectiveness of Stretching on Posterior Shoulder Tightness and Glenohumeral Internal-Rotation Deficit: A Systematic Review of Randomized Controlled Trials. J Sport Rehabil. 2017 Jul;26(4):294-305. doi: 10.1123/jsr.2015-0172. Epub 2016 Aug 24. PMID 27632891
- [Background] Manske R, Wilk KE, Davies G, Ellenbecker T, Reinold M. Glenohumeral motion deficits: friend or foe? Int J Sports Phys Ther. 2013 Oct;8(5):537-53. PMID 24175137
- [Background] Lin DJ, Wong TT, Kazam JK. Shoulder Injuries in the Overhead-Throwing Athlete: Epidemiology, Mechanisms of Injury, and Imaging Findings. Radiology. 2018 Feb;286(2):370-387. doi: 10.1148/radiol.2017170481. PMID 29356641
- [Background] Larrivee S, Balg F, Leonard G, Bedard S, Tousignant M, Boissy P. Wrist-Based Accelerometers and Visual Analog Scales as Outcome Measures for Shoulder Activity During Daily Living in Patients With Rotator Cuff Tendinopathy: Instrument Validation Study. JMIR Rehabil Assist Technol. 2019 Dec 3;6(2):e14468. doi: 10.2196/14468. PMID 31793896
- [Background] Kolber MJ, Vega F, Widmayer K, Cheng MS. The reliability and minimal detectable change of shoulder mobility measurements using a digital inclinometer. Physiother Theory Pract. 2011 Feb;27(2):176-84. doi: 10.3109/09593985.2010.481011. Epub 2010 Aug 8. PMID 20690872
- [Background] Kelly CF, Oliveri Z, Saladino J, Senatore J, Kamat A, Zarour J, Douris PC. The Acute Effect of Tissue Flossing on Pain, Function, and Perception of Movement: A Pilot Study. Int J Exerc Sci. 2023 Jul 1;16(3):855-865. doi: 10.70252/OKAO5505. eCollection 2023. PMID 37637031
- [Background] Keller RA, De Giacomo AF, Neumann JA, Limpisvasti O, Tibone JE. Glenohumeral Internal Rotation Deficit and Risk of Upper Extremity Injury in Overhead Athletes: A Meta-Analysis and Systematic Review. Sports Health. 2018 Mar/Apr;10(2):125-132. doi: 10.1177/1941738118756577. Epub 2018 Jan 30. PMID 29381423
- [Background] Juhan T, Bolia IK, Kang HP, Homere A, Romano R, Tibone JE, Gamradt SC, Weber AE. Injury Epidemiology and Time Lost From Participation in Women's NCAA Division I Indoor Versus Beach Volleyball Players. Orthop J Sports Med. 2021 Apr 27;9(4):23259671211004546. doi: 10.1177/23259671211004546. eCollection 2021 Apr. PMID 33997071
- [Background] Davies GJ, Dickoff-Hoffman S. Neuromuscular testing and rehabilitation of the shoulder complex. J Orthop Sports Phys Ther. 1993 Aug;18(2):449-58. doi: 10.2519/jospt.1993.18.2.449. PMID 8364600
- [Background] Cheatham SW, Nadeau J, Jackson W, Baker R. Effects of Tissue Flossing on Athletic Performance Measures: A Systematic Review. Sports (Basel). 2024 Nov 18;12(11):312. doi: 10.3390/sports12110312. PMID 39590914
- [Background] Challoumas D, Stavrou A, Dimitrakakis G. The volleyball athlete's shoulder: biomechanical adaptations and injury associations. Sports Biomech. 2017 Jun;16(2):220-237. doi: 10.1080/14763141.2016.1222629. Epub 2016 Sep 23. PMID 27659068
- [Background] Cejudo A, Sanchez-Castillo S, Sainz de Baranda P, Gamez JC, Santonja-Medina F. Low Range of Shoulders Horizontal Abduction Predisposes for Shoulder Pain in Competitive Young Swimmers. Front Psychol. 2019 Mar 6;10:478. doi: 10.3389/fpsyg.2019.00478. eCollection 2019. PMID 30894833
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Bonato M, DE Capitani MC, Banfi G. Agility training in volleyball. J Sports Med Phys Fitness. 2022 Jan;62(1):56-64. doi: 10.23736/S0022-4707.21.12084-5. Epub 2021 Feb 22. PMID 33615762
- [Background] Bakshi N, Freehill MT. The Overhead Athletes Shoulder. Sports Med Arthrosc Rev. 2018 Sep;26(3):88-94. doi: 10.1097/JSA.0000000000000200. PMID 30059441
- [Background] Angelopoulos P, Mylonas K, Tsepis E, Billis E, Vaitsis N, Fousekis K. The Effects of Instrument-Assisted Soft Tissue Mobilization, Tissue Flossing, and Kinesiology Taping on Shoulder Functional Capacities in Amateur Athletes. J Sport Rehabil. 2021 Apr 9;30(7):1028-1037. doi: 10.1123/jsr.2020-0200. PMID 33837162